CLINICAL TRIAL: NCT01406782
Title: The Influence of KIR and HLA Genotype on the Response to Rituximab Immunotherapy in Patients With Follicular Lymphoma
Brief Title: DNA Analysis in Influencing Response to Rituximab in Samples From Patients With Follicular Lymphoma Treated on ECOG-E4402
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000706811; ECOG-E4402T3
Record Dates: First submitted 2011-07-29; First posted 2011-08-01 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Rituximab; Gene Expression Profiling; Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Biological: rituximab
Genetic: DNA analysis
Genetic: gene expression analysis
Genetic: polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how well patients will respond to treatment.

PURPOSE: This research study is studying DNA isolated from blood samples to see how well it influences response to rituximab in patients with follicular lymphoma treated on clinical trial ECOG-E4402.

DETAILED DESCRIPTION:
OBJECTIVES:

* To test the influence of killer immunoglobulin-like receptor (KIR) and human lymphocyte antigen (HLA) genotype on response to anti-CD20 antibody lymphoma immunotherapy.

OUTLINE: DNA samples are analyzed for killer immunoglobulin-like receptor (KIR) and human lymphocyte antigen (HLA) genotyping with sequence-specific primers (SSP) by real-time PCR. KIR and HLA typing are analyzed according to KIR-HLA matched vs mismatched, KIR B haplotype content, and the number of inhibitory KIR-HLA pairs. Results are then correlated to each patient's overall response and duration of response to rituximab.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients diagnosed with follicular lymphoma enrolled on ECOG-E4402

  * Treated with single-agent rituximab; the trial compared two different rituximab-dosing strategies - maintenance vs retreatment as needed
* Available germline DNA samples isolated from peripheral blood as well as clinical evaluation of disease status prior to and at initial response to the therapy

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from patients enrolled on E4402 from whom samples were submitted for research
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-12-13 (Actual); Primary Completion 2012-01-13 (Actual); Study Completion 2012-01-13 (Actual)

PRIMARY OUTCOMES:
KIR-HLA genotype predictive of antibody-dependent cell-mediated cytotoxicity (ADCC)-based cancer immunotherapy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Erik Ranheim, MD, PhD, Principal Investigator — University of Wisconsin, Madison